CLINICAL TRIAL: NCT02946307
Title: A Prospective, Multi-center, Randomized, Controlled Clinical Trial, Assessing the Efficacy and Safety of RESTORE Paclitaxel Eluting Balloon Versus RESOLUTE Zotarolimus Eluting Stent for the Treatment of Small Coronary Vessel Disease in Chinese Population With Coronary Heart Disease
Brief Title: Assess the Efficacy and Safety of RESTORE Paclitaxel Eluting Balloon Versus RESOLUTE Zotarolimus Eluting Stent for the Treatment of Small Coronary Vessel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZhuHai Cardionovum Medical Device Co., Ltd. (Industry)
Collaborators: R&G Pharma Studies Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG01W-1102
Record Dates: First submitted 2016-10-24; First posted 2016-10-27 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2018-10

CONDITIONS: Coronary Stenosis
MeSH Terms: conditions — Coronary Stenosis

ARMS (3):
- small vessel cohort:Restore DEB (Experimental): receiving the treatment with Restore DEB（dimeter>2.00 mm） in small vessel cohort
  Interventions: Device: Restore DEB（dimeter>2.00 mm）
- small vessel cohort:Resolute DES (Active Comparator): receiving the treatment with Resolute DES in small vessel cohort
  Interventions: Device: Resolute DES
- very small vessel cohort:Restore DEB (Other): receiving the treatment with Restore DEB（dimeter:2.00 mm）in very small vessel cohort
  Interventions: Device: Restore DEB（dimeter:2.00 mm）

INTERVENTIONS:
Device: Restore DEB（dimeter>2.00 mm）
  Arms: small vessel cohort:Restore DEB
Device: Resolute DES
  Arms: small vessel cohort:Resolute DES
Device: Restore DEB（dimeter:2.00 mm）
  Arms: very small vessel cohort:Restore DEB

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of RESTORE Paclitaxel eluting balloon in the treatment of Chinese patients with coronary heart disease and small vessel lesions in comparison with RESOLUTE Zotarolimus eluting stent.

ELIGIBILITY:
Inclusion Criteria:

Related to the patients:

1. Age ≥18 years old
2. Patients with stable or unstable angina pectoris, or recent myocardial infarction which has been stabilized (occurred over 7 days before enrollment, including non-st segment elevation myocardial infarction(NSTMI) and STMI), or proved asymptomatic regional myocardial ischemia
3. Patients in the small vessel cohort should be suitable for balloon dilation angioplasty or stent implantation, patients in the very small vessel cohort should be suitable for balloon dilation angioplasty.
4. Patients should have sufficient compliance and agree to receive follow-ups in month-1, 6, 9 and 12, and follow-up visit in year-2, 3, 4, and 5. It is required to perform angiography in month-9.
5. Patients should volunteer to participate in this study, and sign the written informed consent form, and understand all risks and benefits in the informed consent document.

   Related to the diseases:
6. Patients with de novo, in situ lesions of small coronary vessels, the length of the lesion should be ≤26mm according to visual inspection. In the small vessel cohort, the diameter of the target lesion should be ≥2.25mm and ≤2.75mm according to visual inspection, and in the very small vessel cohort, the diameter of the target lesion should be ≥2. 00mm and <2.25mm according to visual inspection.
7. The diameter stenosis according to visual inspection before intervention treatment should be ≥70% or ≥50% with the evidence of ischemia.
8. Each patient is allowed to have only one lesion of the target small vessel (2 lesions with the distance ≤10mm and total length ≤26mm which could be treated with the same balloon or stent is considered as one lesion).

Exclusion Criteria:

Related to the patients:

1. Myocardial infarction occurred within 1 week before enrollment.
2. Patients with severe congestive heart failure or New York Heart Association (NYHA) grade IV heart failure
3. Left ventricular ejection fraction (LVEF) <35%
4. Patients who had heart transplantation
5. Patients with severe valvular heart disease
6. The patients had cerebral stroke within 6 months before being included, or have a history of peptic ulcer or gastrointestinal bleeding in the past 6 months, or the patients have a bleeding tendency according to the investigator.
7. Patients with a history of leukopenia (white blood cell count <3×109/L for more than 3 days) or neutropenia (ANC<1000/mm3 for more than 3 days) or thrombocytopenia (platelet <100,000/mm3)
8. Patients with renal insufficiency (eGFR<30ml/min)
9. Patients who are forbidden to use anticoagulation agents or anti-platelet drugs, and unable to tolerate Aspirin or Clopidogrel
10. Patients who are known to be allergic to Paclitaxel or Zotarolimus
11. The patients have a life expectancy of less than 1 year, or it would be difficult to finish follow-ups within 1 year.
12. Pregnant or lactating women, or female patients at a child-bearing age who plan to get pregnant during the period of the study or could not take effective contraceptives
13. The patients are participating in any clinical trials of other drugs or devices before reaching the primary endpoints.
14. Patients who are unsuitable for the study according to the investigator due to other reasons

    Related to the diseases:
15. Patients with total occlusion of the target vessel
16. The patients have severe calcification of the target lesion, and therefore balloon pre-dilation could not be performed successfully.
17. The target lesions are bifurcation lesion with the diameter of the branch vessel >2.00mm.
18. The target lesions are in-stent restenosis.
19. Angiography indicates thrombosis in the target vessel.
20. Complicated with lesions in left main(LM) requiring intervention treatment
21. There are more than 2 non-target lesions which require treatment, or could not be treated with intervention before the target lesion, or the treatment had failed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-08; Primary Completion 2018-12 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
In-segment diameter stenosis(%). | 9 months after the operation.

SECONDARY OUTCOMES:
The success rate of intervention treatment (%),including device success, lesion success and clinical success. | 1-2 days.
In-device diameter stenosis (%) of the target lesion. | 9 months after the operation.
cardiac death. | in month-1, 6, 9, 12 and year-2, 3, 4, 5.
myocardial infarction related to the target vessel. | in month-1, 6, 9, 12 and year-2, 3, 4, 5.
target lesion revascularization driven by ischemia. | in month-1, 6, 9, 12 and year-2, 3, 4, 5.
all-cause death | in month-1, 6, 9, 12 and year-2, 3, 4, 5.
myocardial infarction | in month-1, 6, 9, 12 and year-2, 3, 4, 5.
any target lesion revascularization | in month-1, 6, 9, 12 and year-2, 3, 4, 5.
acute thrombosis | in month-1, 6, 9, 12 and year-2, 3, 4, 5
sub-acute thrombosis | in month-1, 6, 9, 12 and year-2, 3, 4, 5
end-stage thrombosis | in month-1, 6, 9, 12 and year-2, 3, 4, 5
delayed thrombosis | in month-1, 6, 9, 12 and year-2, 3, 4, 5

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, Master, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (12):
- China (12):
  - Beijing Anzhen Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Fuwai Hospital, CAMS&PUMC, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital, The Affiliated Hospital of Najing University Medical School, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Tangdu Hospital, Xi'an, Shaanxi
  - Tianjin 4th Centre Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Li L, Guan C, Meng S, Bai Y, Zhang Z, Zou K, Ruan Y, Cao X, Jia R, Guo C, Escaned J, Jin Z, Xu B. Short- and long-term functional results following drug-coated balloons versus drug- eluting stents in small coronary vessels: The RESTORE quantitative flow ratio study. Int J Cardiol. 2021 Mar 15;327:45-51. doi: 10.1016/j.ijcard.2020.11.035. Epub 2020 Nov 21. PMID 33227335
- [Derived] Tang Y, Qiao S, Su X, Chen Y, Jin Z, Chen H, Xu B, Kong X, Pang W, Liu Y, Yu Z, Li X, Li H, Zhao Y, Wang Y, Li W, Tian J, Guan C, Xu B, Gao R; RESTORE SVD China Investigators. Drug-Coated Balloon Versus Drug-Eluting Stent for Small-Vessel Disease: The RESTORE SVD China Randomized Trial. JACC Cardiovasc Interv. 2018 Dec 10;11(23):2381-2392. doi: 10.1016/j.jcin.2018.09.009. PMID 30522667